CLINICAL TRIAL: NCT05361148
Title: Long-term Health After Severe Acute Malnutrition in Children and Adults: the Role of the Pancreas
Acronym: SAMPA
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Newcastle University, UK (Unknown); University of Copenhagen (Other); National Institute for Medical Research, Tanzania (Other Government); Nutrition Centre of the Philippines (Unknown); University Teaching Hospital, Lusaka, Zambia (Other); Delhi University (Other)
Responsible Party: Sponsor
Other Study IDs: EPPHZU29
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-10

CONDITIONS: Pancreas Atrophy; Diabetes; Malnutrition
Keywords: diabetes; exocrine pancreas; endocrine pancreas; malnutrition
MeSH Terms: conditions — Diabetes Mellitus; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma feces urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- DIVIDS (Delhi Infant Vitamin D Supplementation) study, India: The DIVIDS cohort were born low birth weight (LBW, <2.5 kg) at term in 2007-2010. They had monthly follow-up until 6m then at 5 and 11 years. Anthropometry was collected at all visits, body composition in the 5 and 11 years, and blood samples at 6 months and 5 and 11 years. For SAMPA, the DIVIDS cohort acts as a positive control since we expect adverse long-term non-communicable disease consequences of being born LBW.
  Sample numbers at previous follow-ups and expected:
  * Birth: 2079 total, all LBW
  * Age 5 y: 911 total, 764 (84%) BMIZ>-2, 138 (15%) BMIZ -2 to -3, 9 (1%) BMIZ<-3
  * Age 11 y (ongoing): 647 total, 482 (75%) BMIZ>-2, 117 (18%) BMIZ -2 to -3, 48 (7%) BMIZ<-3
  * Expected for SAMPA: 800 total
  Interventions: Other: no interventions will be used
- SAM (Severe Acute Malnutrition) Lusaka: This group comprises children with or without prior MALN in early childhood. Some are from a study which identified 1195 children with MALN (mean age 16 months, 11.6% HIV-infected) in a house-to-house survey in a low-income area, Misisi, Lusaka in 2009. Some children are from a study of body composition and indicators of chronic diseases (HbA1c, lipids); 100 were hospitalised with MALN when < 2 years and 76 are never-malnourished neighbourhood controls.
  Sample numbers at previous follow-ups and expected:
  * Age < 2 y: 400 total, 200 WHZ<-3, 200 well-nourished
  * Age 9 y: 186 total, 110 previous MALN, 76 no MALN; currently 17 (9%) BMIZ <-2
  * Expected for SAMPA: 400 total
  Interventions: Other: no interventions will be used
- CICADA (Chronic Infections, Co-morbidities and Diabetes in Africa), Mwanza, Tanzania: The CICADA cohort comprises HIV-infected and uninfected recruited since 2010. CICADA involved 3 annual visits for data on HbA1c, OGTT, insulin, anthropometry, body composition, and diabetes lifestyle risk factors. CICADA has the most detailed longitudinal diabetes data of the project cohorts, archived fasting samples, and are the oldest so have had longer to develop diabetes; therefore, this cohort will be used for the in-depth and longitudinal components (hypotheses 3 and 4).
  Sample numbers at previous follow-ups and expected:
  * 12 y prior: 447 total, 300 (67%) BMI > 18.5 kg/m2, 74 (17%) BMI 17 to 18.5 kg/m2 73 (16%) BMI <17 kg/m2
  * 10 y prior: 704 total, 304 (43%) BMI 17 to 18.5 kg/m2, 400 (57%) BMI<17 kg/m2
  * 3 y prior: 1947 total, 1519 (78%) BMI > 18.5 kg/m2, 275 (14%) BMI 17 to18.5 kg/m2, 152 (8%) BMI <17 kg/m2
  * Expected for SAMPA: 1200 total
  Interventions: Other: no interventions will be used
- NUSTART Lusaka: We will trace and recruit 200 previously malnourished HIV-infected adults from the NUSTART Lusaka participants plus 100 non-HIV-infected neighbourhood controls to the SAMPA study. As for NUSTART Mwanza, there was a high mortality rate during the first 12 weeks of ART.
  Sample numbers at previous follow-ups and expected:
  * 10 y prior: 1111 total, 437 (39%) BMI 17 to 18.5 kg/m2, 674 (61%) BMI<17 kg/m2
  * Expected for SAMPA: 300 total
  Interventions: Other: no interventions will be used
- St-ATT (Starting Anti-TB Treatment) Cohort, Philippines: Between Aug 2018 and Feb 2020, the St-ATT cohort recruited 900 adults within 5 days of starting a new 6 or 9 month anti-TB regimen in three provinces: Cebu, Negros Occidental and Metro Manila, encompassing urban, peri-urban and rural populations. 17% had HbA1c >=7.0% (probable diabetes in TB) with an additional 30% with HbA1c 5.8%-7.0% ('prediabetes'/mild TB-induced hyperglycaemia). Post-treatment follow-up is ongoing. This cohort will be involved in in-depth analyses for hypothesis 3.
  Sample numbers at previous follow-ups and expected:
  * 1-2 y prior: 900 total, 495 BMI >18.5 kg/m2, 189 (21%) BMI 17.0 -18.5 kg/m2, 216 (24%) BMI <17 kg/m2
  * Expected for SAMPA: 600 total
  Interventions: Other: no interventions will be used
- CLHNS (Cebu Longitudinal Health and Nutrition Survey), Philippines: The cohort was recruited in 1983-84. Since the original follow-up to age 2 years, there have been 8 follow-up surveys including in 2019 when 1300, ~40% of the initial cohort, were available. Loss from the cohort over time is mostly from out-migration and those remaining are more rural and of lower socioeconomic status. In follow-up surveys, data collection included: anthropometry, diet (24-hr recall), health history, blood pressure and other chronic disease risk factors, school achievement, and, for older ages, reproductive history. This cohort represents our longest follow-up of MALN diagnosed by anthropometry resulting primarily from poor nutrition, not specific severe infections.
  Sample numbers at previous follow-ups and expected:
  * Birth: 28 LBW of the 144 with childhood MALN
  * Age < 2 y: of 420 total to be included, 144 (34%) WHZ<-3
  * Expected for SAMPA: 420 total
  Interventions: Other: no interventions will be used

INTERVENTIONS:
Other: no interventions will be used — This is a cohort study with no interventions.

SUMMARY:
Whilst there is an increasing prevalence of overweight and obesity worldwide, malnutrition remains common. In addition, malnutrition, overweight, and infections often interact. The consequences of malnutrition after birth are little studied. Severe acute malnutrition in childhood remains common in Africa and Asia and many adult patients with tuberculosis or HIV, diseases which are common in Africa and Asia, may become malnourished. The investigators are interested in diabetes, which in Africa and Asia affects people at younger age and lower weight than in Europe. There is evidence that severe postnatal malnutrition increases the risk of later diabetes but the evidence is piecemeal and there is little information as to the mechanisms involved. It is thus difficult to determine what treatments or preventative strategies are appropriate.

The investigators wish to focus on the pancreas which is a key organ in digestion and metabolic processes, especially in relation to diabetes. They will investigate pancreas size, microscopic structure, hormone and digestive enzyme production, and the body's response to these hormones among groups of people in Tanzania, Zambia, India and the Philippines. These groups have participated in the research team's previous studies of malnutrition and were malnourished before birth, as children, or as adults. They now live in places with a wide range of access to foods high in fat and sugar which could affect their risk of diabetes. The investigators will compare their pancreas function to that of never-malnourished controls at each site. The investigators will use advanced statistical methods to understand the links between early malnutrition and later diabetes, taking into account the factors often associated with diabetes such as age, current overweight and infection.

Even if the investigators find no important link between early malnutrition and later diabetes, the research will lead to improved understanding of the long-term consequences of malnutrition and the presentation and underlying metabolism of diabetes in Africa and Asia. Thus, the project will lead to improved health care for both malnourished and diabetic people.

DETAILED DESCRIPTION:
Prenatal growth retardation is associated with increased risk of adult chronic non-communicable diseases (NCDs) including diabetes. However, there is limited information regarding how postnatal malnutrition, in childhood or adulthood, affects these risks. The question of long-term effects of postnatal malnutrition is of increasing importance, because, with improved care, more children survive severe acute malnutrition and, amongst adults, drug treatments for infections, e.g. HIV and tuberculosis which frequently cause or are associated with malnutrition (MALN), have improved patient survival. Our project will focus on the role of the pancreas in the long-term consequences of MALN since both its endocrine and exocrine functions are critical for nutrition and NCDs. There is evidence that pancreatic functions may not recover fully after childhood or adult MALN and that the phenotype of diabetes in countries with prevalent MALN differs from that in high-income countries.

Overall hypothesis:

Severe malnutrition (MALN) at any age has medium- and long-term detrimental effects on endocrine and exocrine pancreatic function and structure.

Study design and population: Cross-sectional observational study recruiting a total of 3700 participants from previous/ongoing observational cohorts in: Zambia (1 adult (N=300) and 1 adolescent cohort (N=180)), Tanzania (1 adult cohort (N=1400)), Philippines (2 adult cohorts N=600/N=420), India (1 adolescent low birth weight cohort N=800))

Specific objective 1: To determine if MALN earlier in life is associated with abnormalities of pancreas structure and function.

Hypothesis 1: Prior MALN is associated with later abnormal pancreatic structure and endocrine and exocrine function.

Approach: The investigators will follow up individuals from the above cohorts in which there are participants, all now adolescents or adults, who suffered from MALN at different stages earlier in life as well as age- and sex-matched individuals who have never been malnourished as a comparison. The researchers will assess in those with and without prior MALN:

1. blood glucose, insulin and C-peptide during an oral glucose tolerance test (OGTT)
2. haemoglobin A1c (HbA1c)
3. faecal elastase and plasma lipase as exocrine pancreas markers
4. pancreas size and architecture using ultrasound and computed tomography (CT) (subset)

Specific objective 2: To investigate whether pancreatic abnormalities in participants with prior MALN and diabetes are compatible with a previously prescribed entity of fibro-calculous diabetes.

Hypothesis 2: Prior MALN is associated with pancreatic calcifications and is common in those with diabetes.

Approach: The investigators will conduct CT scans to investigate pancreatic calcification among non-pregnant adult study participants.

Specific objective 3: To investigate the relative importance of decreased insulin production or increased insulin resistance in MALN associated with concurrent infections in African and Asian adult populations.

Hypothesis 3: The abnormal glucose regulation seen after MALN and infection is associated with relative insulin deficiency with or without insulin resistance.

Approach: This hypothesis will be investigated within the Tanzanian cohort and one Filipino adult cohort, both of whom had MALN associated with infection. 20 men and 20 women will be selected from each of two groups (MALN and non-MALN) in each cohort based on whether or not in our prior research they were recorded as experiencing MALN. In these participants the investigators will:

1. Measure in blood samples collected at 0, 15, 30, 45, 60, 90 and 120 minutes during an OGTT: glucose, insulin, C-peptide (all time points), the incretins gastric inhibitory polypeptide (GIP) and glucagon-like peptide-1 (GLP-1) and glucagon at 0, 30, 60, 90 and 120 minutes, and proinsulin and trypsinogen at baseline only;
2. Conduct intravenous glucose tolerance tests (IVGTT) and measure in blood samples collected at -10, -1, 2, 4, 6, 8, 10 minutes: glucose, insulin, and C-peptide.

Specific objective 4: To investigate whether a prior abnormal pro-insulin / insulin ratio is associated with diabetes in adults infected with HIV or previously with tuberculosis.

Hypothesis 4: An abnormal pro-insulin/insulin ratio is associated with later development of diabetes in adults who had MALN and infection.

Approach: For participants from the CICADA, Tanzania, cohort the reasearch team has fasting plasma samples stored from prior follow-ups up to 10 years earlier. Glucose has already been measured in these samples as well as insulin in some samples. The investigators will measure insulin in the remaining stored samples and proinsulin in all to investigate whether prior proinsulin / insulin ratio is associated with subsequent diabetes.

ELIGIBILITY:
Inclusion Criteria:

* member of one of the 6 included cohorts
* informed consent (for children, informed assent and consent of guardian)

Exclusion Criteria:

* lack of consent
* pregnant women and chidlren will be excluded from CT scans and interavenous glucose tolerance tests

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population are members of one of the 6 cohorts described above
Sampling Method: Non-Probability Sample
Enrollment: 2305 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Pancreas endocrine function | 1 year
  Mathematical modelling of blood glucose, insulin and C-peptide at 3 (for children) or 7 (for adults) times during a 120 minute oral glucose tolerance test (OGTT) to determine first and second phase insulin release and insulin resistance
Pancreas exocrine function | 1 year
  faecal elastase and plasma lipase

SECONDARY OUTCOMES:
Pancreas size and structure | 1 year
  pancreas size and architecture using ultrasound and computed tomography (CT) (subset)
pancreatic calcification | 1 year
  calcification determined by CT scan (subset)
Hemoglobin A1c | 1 year
  blood HbA1c as diabetes marker
insulin production and insulin resistance (in-depth study in a subset) | 1 year
  Mathematical modelling of data from analytes from an intravenous glucose tolerance tests (IVGTT) in a subset and measure in blood samples collected at -10, -1, 2, 4, 6, 8, 10 minutes: glucose, insulin, and C-peptide Combined results will be used to indicate first and second phase insulin production and insulin resistance.
gastrointestinal contribution to glucose metabolism and diabetes | 1 year
  Incretins (gastric inhibitory polypeptide (GIP) and glucagon-like peptide-1 (GLP-1)) and glucagon at 0, 30, 60, 90 and 120 minutes during an OGTT
Proinsulin | 1 year
  proinsulin in baseline samples before OGTT
abnormal prior pro-insulin/insulin ratio and diabetes (subset) | 1 year
  From CICADA cohort, measurement of pro-insulin and insulin in samples collected 4 years previously and compare with current diabetes by OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Filteau, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (4):
- Institute of Home Economics Delhi University, Delhi, India
- Nutrition Centre of the Philippines, Cebu City, Philippines
- National Institute for Medical Research, Mwanza, Tanzania
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No
Data can be made available for bona fide research conducted under the conditions of the original ethical approvals. Interested researchers should contact the principal investigator.